CLINICAL TRIAL: NCT06800326
Title: Diagnostic Concordance of MR Enterography and Ultrasound for Treatment Response Assessment in Crohn's Disease (MANTRA): a Multicentre, Non-randomised, Multiple-arm, Prospective Cohort Comparison Study
Brief Title: Diagnostic Concordance of MR Enterography and Ultrasound for Treatment Response Assessment in Crohn's Disease (MANTRA)
Status: Recruiting | Type: Observational
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: 172896
Record Dates: First submitted 2024-07-29; First posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ultrasound Scan: An additional follow up IUS i.e. all participants undergo both a follow up MRE and IUS, with no participant randomisation. The cohort under US would have had an MRE as part of their standard of care.
  Interventions: Diagnostic Test: Ultrasound; Diagnostic Test: MRE Scan
- MRE Scan: An additional follow up MRE i.e. all participants undergo both a follow up MRE and IUS, with no participant randomisation. The cohort under MRE would have had an IUS as part of their standard of care.
  Interventions: Diagnostic Test: Ultrasound; Diagnostic Test: MRE Scan

INTERVENTIONS:
Diagnostic Test: Ultrasound — Participants will have either an ultrasound or magnetic resonance imaging, depending on what scan they have had as part of their standard of care.
Diagnostic Test: MRE Scan — Participants will have either an ultrasound or magnetic resonance imaging, depending on what scan they have had as part of their standard of care.

SUMMARY:
Crohn's disease is a lifelong condition resulting in inflammation of the bowel. Treatment with powerful drugs aim to reduce inflammation by suppressing the immune system. It is important to regularly assess if the drugs are effective, so they can be stopped or changed if not.

There are several ways doctors assess if the medication is effective as just relying on how the patient feels is not sufficient. Blood and stool tests looking for inflammation are useful but have limitations. Looking into the bowel using endoscopy is effective but very invasive. Medical imaging notably MR Enterography (MRE), a type of MRI scan, and intestinal ultrasound (IUS) visualise the bowel, and are safe, non-invasive and generally well tolerated tests frequently used in the NHS to assess how well treatment is working.

There is however wide variation in which imaging test is selected without clear guidance. The investigators currently do not know if one is better in assessing response to treatment, and if they can be used interchangeably.

The proposed study will investigate this question to guide the future care of Crohn's disease patients. The investigators will recruit patients having follow up imaging tests to assess their treatment and ask them to undergo both MRE and IUS. Radiologists will interpret the MRE and IUS, unaware of the findings of the other test, and state if the disease is improving or not. The doctors looking after the patient will then look at all available information e.g. symptoms, blood/stool tests, colonoscopy, and decide if the patient is the same, worse or better on the medication. This decision will be used to establish how accurate MRE and IUS are in assessing response, how often they agree and if they can be used interchangeably in the future, for example based on patient preference or availability at the hospital.

DETAILED DESCRIPTION:
Imaging, typically with MR enterography (MRE) and/or Intestinal Ultrasound (IUS), is central in the follow up of Crohn's disease patients to assess treatment response to powerful immunosuppressive therapy. Practice varies widely on which imaging modality is selected and/or available and if they are used in isolation or interchangeably. There is currently no set guidance and practice varies widely.

We know that both MRE and IUS are accurate for diagnosing and staging Crohn's disease, although patients generally prefer IUS if it is of comparable accuracy. We however do not understand if MRE and IUS can be used interchangeably for treatment response assessment. Such uncertainty can impede patients and clinical teams in making informed management decisions.

Currently, IUS provision is sparse with no formal training programme, leading to a heavy bias for MRE. This approach is more costly, less tolerable to patients, adds pressure to already overloaded MRI workflows, and less environmentally sustainable. The current study may support the drive for comprehensive provision of both MRE and IUS services and training.

Currently, the literature is very limited and largely comprised of small single centre studies (most less than 50 patients), using inconsistent imaging definitions of treatment response, highly varied reference standards and differing follow up intervals. There are several MRE and IUS scores for objective disease assessment which remain to be fully validated for response and their respective agreement is not fully understood.

Ultimately, a major outstanding research question is not if investigators should use MRE or IUS, but rather, when investigators should use them in the management of individual patients. Accordingly, the European Society of Gastrointestinal and Abdominal Radiology (ESGAR) and the James Lind Alliance/Crohn's & Colitis UK identify the current study topic as a key research priority.

The proposed prospective study will be the largest to date to investigate the accuracy of MRE and IUS for classification of treatment response against an expert consensus panel, their agreement in response assessment.

ELIGIBILITY:
Inclusion Criteria:

* Small bowel or colonic Crohn's disease
* 16 years or older
* Baseline/pre-treatment MR Enterography or Intestinal Ultrasound already performed as part of standard clinical care
* Follow up MR Enterography or Intestinal Ultrasound requested to assess treatment response within 15 months of baseline/ pre-treatment imaging

Exclusion Criteria:

* Interval resection of diseased segment(s)
* Inability to achieve informed consent
* Pregnancy
* Any contraindication/ intolerance to MRI

Ages: 16 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be male and female from 16 years and above who have small bowel or colonic Crohn's disease.
Sampling Method: Non-Probability Sample
Enrollment: 155 (Estimated)
Dates: Start 2024-10-04 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Measure | 18 months
  The primary outcome will measure the difference in the percentage correct treatment response classification using MR Enterography (MRE) and Intestinal Ultrasound (IUS), against a multidisciplinary consensus panel reference standard.

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Taylor, Principal Investigator — UCLH
Locations (1):
- University College London Hospitals, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Radford SJ, Taylor S, Moran G. Ultrasound use to assess Crohn's disease in the UK: a survey of British Society of Gastroenterology Inflammatory Bowel Disease Group members. Frontline Gastroenterol. 2022 Jan 18;13(6):471-476. doi: 10.1136/flgastro-2021-102065. eCollection 2022. PMID 36250164
- [Result] Taylor SA, Mallett S, Bhatnagar G, Baldwin-Cleland R, Bloom S, Gupta A, Hamlin PJ, Hart AL, Higginson A, Jacobs I, McCartney S, Miles A, Murray CD, Plumb AA, Pollok RC, Punwani S, Quinn L, Rodriguez-Justo M, Shabir Z, Slater A, Tolan D, Travis S, Windsor A, Wylie P, Zealley I, Halligan S; METRIC study investigators. Diagnostic accuracy of magnetic resonance enterography and small bowel ultrasound for the extent and activity of newly diagnosed and relapsed Crohn's disease (METRIC): a multicentre trial. Lancet Gastroenterol Hepatol. 2018 Aug;3(8):548-558. doi: 10.1016/S2468-1253(18)30161-4. Epub 2018 Jun 18. PMID 29914843
- [Result] Rimola J, Torres J, Kumar S, Taylor SA, Kucharzik T. Recent advances in clinical practice: advances in cross-sectional imaging in inflammatory bowel disease. Gut. 2022 Dec;71(12):2587-2597. doi: 10.1136/gutjnl-2021-326562. Epub 2022 Aug 4. PMID 35927032
- [Result] Novak KL, Nylund K, Maaser C, Petersen F, Kucharzik T, Lu C, Allocca M, Maconi G, de Voogd F, Christensen B, Vaughan R, Palmela C, Carter D, Wilkens R. Expert Consensus on Optimal Acquisition and Development of the International Bowel Ultrasound Segmental Activity Score [IBUS-SAS]: A Reliability and Inter-rater Variability Study on Intestinal Ultrasonography in Crohn's Disease. J Crohns Colitis. 2021 Apr 6;15(4):609-616. doi: 10.1093/ecco-jcc/jjaa216. PMID 33098642